CLINICAL TRIAL: NCT06425419
Title: The Safety and Efficacy of Intravitreal Topotecan for the Treatment of Proliferative Vitreoretinopathy
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Leo Am Kim, M.D., Associate Professor of Ophthalmology, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023P002259
Record Dates: First submitted 2024-01-09; First posted 2024-05-22 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Proliferative Vitreoretinopathy; Proliferative Vitreo-Retinopathy; Rhegmatogenous Retinal Detachment
MeSH Terms: conditions — Vitreoretinopathy, Proliferative | interventions — Topotecan

STUDY DESIGN:
Intervention Model Description: Half of the patients will receive intravitreal topotecan at the time of surgery. Randomization will be done based on a computer-generated list that would randomly allocate each of the 50 participants to being either in the treatment arm or in the control arm, in a particular order. Results will be printed on a card put in sealed envelopes that would be given to each research subject based on the allocation order given by that computer-generated list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Participants who received intravitreal topotecan (Experimental): These are the patients who will be receiving intravitreally 20 micrograms of topotecan in a 1cc syringe during surgery, at the post-operative day 7 and at the post-operative day 28.
  Interventions: Drug: Topotecan
- Participants who did not received intravitreal topotecan (No Intervention): These patients will not be receiving any intervention.

INTERVENTIONS:
Drug: Topotecan — 20 micrograms of intravitreal topotecan given in a 1 cc tuberculin syringe at a concentration of 20 mcg/20mcL.
  Other Names: Hycamtin
  Arms: Participants who received intravitreal topotecan

SUMMARY:
The goal of this clinical trial is to evaluate the safety and efficacy of intravitreal topotecan for the treatment of patients with rhegmatogenous retinal detachment due to proliferative vitreoretinopathy (PVR) or resulting from an open globe injury, and compare the outcomes to those who do no receive intravitreal topotecan. The main objectives it aims to achieve are:

* to study the safety profile of intravitreal topotecan in the treatment of PVR
* to evaluate the efficacy of intravitreal topotecan in treating PVR.

Post-consent, participants will:

* undergo vitrectomy (with or without scleral buckle) as part of standard treatment for retinal detachment.
* receive intravitreal topotecan at the time of surgery, post-operative day 7 and post-operative day 28 (if randomized to receive the medication)
* come in at post-operative day 1, 7, 28, 56, 84, 126 and 168 to undergo a complete ophthalmic exam along with a fundus photography and optical coherence tomography of the macula, have their intraocular pressure and visual acuity measured and their adverse events monitored, if any.

Researchers will compare participants who receive intravitreal topotecan for PVR to those who do not to see if there is a significant variability in recurrence of retinal detachment, rate of retinal reattachment and PVR grade 6 months after surgery.

DETAILED DESCRIPTION:
Rhegmatogenous retinal detachment (RRD) is an acute, sight-threatening condition that occurs after separation of the neurosensory retina from the underlying retinal pigment epithelium (RPE) due to the presence of a retinal break. Proliferative vitreoretinopathy (PVR) represents growth of ectopic fibrocellular growth on the surface of, within and underneath the retina. PVR is hypothesized to occur secondary to the migration of RPE cells to the peri-retina, leading to a mesenchymal transition into contractile myofibroblasts. PVR affects 5-10% of RRDs and is the most common cause of surgical failure in RRD.

Given that PVR involves a pro-inflammatory and pro-fibrotic cellular response, adjuvants such as corticosteroids and antimetabolites such as 5-fluorouracil have been attempted in the treatment of this condition. Overall, the efficacy results of these treatments have been mixed, and no standard of care adjuvant therapy has emerged.

Topotecan is a chemotherapeutic agent that acts as a topoisomerase inhibitor. It is most commonly administered intravitreally for patients with refractory or recurrent vitreous seeds from retinoblastoma, and shows high efficacy in this setting. At the same time, intravitreal topotecan administered at doses of 5-30µg has been associated with no ocular or systemic complications or adverse electroretinogram changes. To the best of available knowledge, topotecan has not been administered for the treatment of proliferative vitreoretinopathy. Topotecan has anti-inflammatory, anti-proliferative and anti-fibrotic activity that is hypothesized to exhibit high efficacy for the treatment of PVR. In this study, the efficacy and safety of intravitreal topotecan for the treatment of PVR will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 18 years old
* Patients presenting with retinal detachment due with PVR (grade C or higher) or retinal detachment associated with open globe trauma
* Patients undergoing vitrectomy or vitrectomy with scleral buckle as part of standard care.

Exclusion Criteria:

* Patient unable to give consent
* Patient unable to follow-up
* Females of childbearing age who are pregnant at the time of recruitment. A pregnancy test will be done to all women of ages 18-55 prior to surgery to ensure they are not pregnant at the time of recruitment.
* Patients with a history of tractional or exudative retinal detachment.
* Patients with other planned ocular surgery following PPV
* Active or chronic or recurrent uncontrolled ocular or systemic disease
* Active or history of chronic or recurrent inflammatory eye disease
* Diagnosis of severe nonproliferative or proliferative diabetic retinopathy or vasoproliferative disease in the operative eye
* Signs of ocular infection at presentation in either eye
* Known or suspected sensitivity or allergy to any of the medications used in the operation or postoperatively
* No Light Perception vision in the operative eye
* Failure to achieve intraoperative reattachment
* Patient with silicone oil instilled in the operative eye at time of presentation

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence of rhegmatogenous retinal detachment secondary to PVR | 6 months after initial surgery, or last follow-up visit available
  Investigators will be evaluating whether participant develop a recurrent retinal detachment throughout their follow up after their initial surgery.

SECONDARY OUTCOMES:
Best corrected visual acuity (BCVA) | at the pre-operative assessment, and post-operative day1, 7, 28, 56, 84, 126, 168
  Investigators will be measuring the BCVA of participants throughout their follow up and see if they notice any change from surgery time to final follow up
Variation of PVR grade | at the pre-operative assessment, and post-operative day1, 7, 28, 56, 84, 126, 168
  Investigators will be doing a dilated fundus exam and taking fundus photographies for all participants throughout their follow up time to see if the grade of the PVR changes over time. PVR grade goes from grade A to grade C-Anterior to equator/ C-Posterior to equator (grade C being worse than grade A)
Retinal reattachment rate at month 6 or last follow up | at post-operative day 168 (or last follow-up visit available if the participant did not show up at post-operative day 168)
  Investigators will be doing a dilated fundus exam and taking fundus photographies for all participants throughout their follow up time to see if the retinal reattaches (whether completely or partially) after surgery
Recurrence of rhegmatogenous retinal detachment due to any cause | at the pre-operative assessment, and post-operative day1, 7, 28, 56, 84, 126, 168
  Investigators will be measuring the BCVA of participants throughout their follow up and see if they notice any change from surgery time to final follow up
Number of participants and type of intraoperative or postoperative complications | at time of surgery, and each follow up visit (post-operative day1, 7, 28, 56, 84, 126, 168)
  Any adverse event will be noted during surgery, and at each follow up visit for each participant if applicable.

OTHER OUTCOMES:
Optical coherence tomography (OCT) of the macula | at the pre-operative assessment, and post-operative day1, 7, 28, 56, 84, 126, 168
  an OCT of the macula will be taken to evaluate for any retinal changes throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Leo Kim, MD, PhD, Principal Investigator — Massachusetts Eye and Ear

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ohman T, Gawriyski L, Miettinen S, Varjosalo M, Loukovaara S. Molecular pathogenesis of rhegmatogenous retinal detachment. Sci Rep. 2021 Jan 13;11(1):966. doi: 10.1038/s41598-020-80005-w. PMID 33441730
- [Background] Mysore Y, Del Amo EM, Loukovaara S, Hagstrom M, Urtti A, Kauppinen A. Statins for the prevention of proliferative vitreoretinopathy: cellular responses in cultured cells and clinical statin concentrations in the vitreous. Sci Rep. 2021 Jan 13;11(1):980. doi: 10.1038/s41598-020-80127-1. PMID 33441813
- [Background] Claes C, Lafeta AP. Proliferative vitreoretinopathy. Dev Ophthalmol. 2014;54:188-95. doi: 10.1159/000360466. Epub 2014 Aug 26. PMID 25196769
- [Background] Pastor JC, de la Rua ER, Martin F. Proliferative vitreoretinopathy: risk factors and pathobiology. Prog Retin Eye Res. 2002 Jan;21(1):127-44. doi: 10.1016/s1350-9462(01)00023-4. PMID 11906814
- [Background] Sadaka A, Giuliari GP. Proliferative vitreoretinopathy: current and emerging treatments. Clin Ophthalmol. 2012;6:1325-33. doi: 10.2147/OPTH.S27896. Epub 2012 Aug 14. PMID 22942638
- [Background] Rao R, Honavar SG, Sharma V, Reddy VAP. Intravitreal topotecan in the management of refractory and recurrent vitreous seeds in retinoblastoma. Br J Ophthalmol. 2018 Apr;102(4):490-495. doi: 10.1136/bjophthalmol-2017-310641. Epub 2017 Aug 26. PMID 28844050
- [Background] Bogan CM, Kaczmarek JV, Pierce JM, Chen SC, Boyd KL, Calcutt MW, Bridges TM, Lindsley CW, Nadelmann JB, Liao A, Hsieh T, Abramson DH, Francis JH, Friedman DL, Richmond A, Daniels AB. Evaluation of intravitreal topotecan dose levels, toxicity and efficacy for retinoblastoma vitreous seeds: a preclinical and clinical study. Br J Ophthalmol. 2022 Feb;106(2):288-296. doi: 10.1136/bjophthalmol-2020-318529. Epub 2021 May 10. PMID 33972235
- [Background] Nadelmann J, Francis JH, Brodie SE, Muca E, Abramson DH. Is intravitreal topotecan toxic to retinal function? Br J Ophthalmol. 2021 Jul;105(7):1016-1018. doi: 10.1136/bjophthalmol-2020-316588. Epub 2020 Jul 14. PMID 32665221
- [Background] Ghassemi F, Shields CL, Ghadimi H, Khodabandeh A, Roohipoor R. Combined intravitreal melphalan and topotecan for refractory or recurrent vitreous seeding from retinoblastoma. JAMA Ophthalmol. 2014 Aug;132(8):936-41. doi: 10.1001/jamaophthalmol.2014.414. PMID 24789622
- [Background] Cepeda MS, Boston R, Farrar JT, Strom BL. Comparison of logistic regression versus propensity score when the number of events is low and there are multiple confounders. Am J Epidemiol. 2003 Aug 1;158(3):280-7. doi: 10.1093/aje/kwg115. PMID 12882951
- [Background] Kim J, Shin W. How to do random allocation (randomization). Clin Orthop Surg. 2014 Mar;6(1):103-9. doi: 10.4055/cios.2014.6.1.103. Epub 2014 Feb 14. PMID 24605197
- [Background] Machemer R, Aaberg TM, Freeman HM, Irvine AR, Lean JS, Michels RM. An updated classification of retinal detachment with proliferative vitreoretinopathy. Am J Ophthalmol. 1991 Aug 15;112(2):159-65. doi: 10.1016/s0002-9394(14)76695-4. PMID 1867299